CLINICAL TRIAL: NCT03599973
Title: Corrélation Entre la Longueur de jeûne et la réponse au Remplissage Vasculaire évaluée Par Des Mesures répétées de l'ITV.
Brief Title: Correlation Between Duration of Fasting and Response to Fluid Replenishment, Evaluated With Repeated Measures of VTI.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ErasmeVTI2018
Record Dates: First submitted 2018-04-13; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-06

CONDITIONS: Fluid and Electrolyte Imbalance; Fluid Therapy
Keywords: Rehydration Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patient (Other): One-arm study, where all patients are given the same standard fluidotherapy and anesthetic conditions to compare measures of Aortic VTI before and after the IV fluid.
  Interventions: Other: Plasmalyte A Viaflo

INTERVENTIONS:
Other: Plasmalyte A Viaflo — Fluid therapy to be given according to the principle of 4-2-1 (4 ml of crystalloid fluid for each of the first 10 kg of weight (0-10 kg), 2 ml of crystalloid fluid for each of the second 10 kg of weight (11-20 kg) and 1 ml of crystalloid fluid for each kg of weight over 20.

SUMMARY:
The investigators will study the correlation between the lenght of the fasting before surgery and the need to replenish with intra-venous fluids in children, evaluated with 3 measures of the aortic Integral Time Velocity with transthoracic echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 3 and 6 years with a normal ponderal evolution.
* Children with good general status (ASA 1)
* Children whose parents have given the informed authorization to do the study.
* Children seen in the consultation of anesthesiology.
* Children programed to have ambulatory surgery (Amygdalectomy, dental care, dental extraction).

Exclusion Criteria:

* Children with more than 6 years of age.
* Children whose parents didn't agree with the study.
* Children enrolled in another study on the 3 months before.
* Children with hearth or lung conditions.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2018-08-15 (Estimated); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
Aortic VTI change | From baseline analysis (t=5 min after anesthesia induction), to the end of fluid therapy (t=20 min).
  Transthoracic echocardiography measures of the Time-Speed Interval in the aortic valve before fluid therapy (baseline) and after fluid therapy (20 ml/kg in 15 minutes).

SECONDARY OUTCOMES:
Blood pressure change | From baseline analysis (t=5 min after anesthesia induction), to the end of fluid therapy (t=20 min).
  Analysis of the variation of Mean Arterial Blood pressure with fluid therapy
Legs-up maneuver | From baseline analysis (t=5 min after anesthesia induction), to the end of legs-up maneuver (t = +/- 10 min).
  Analysis of the variation of Mean Arterial Blood pressure with the legs up maneuver
Post-operative nausea and vomiting | From arrival at PACU (end of surgery) until discharge from PACU (tipically after 1 to 2 hours after the arrival to the PACU)
  Comparisson of the incidence of post-operative nausea and vomiting in the fluid respondeurs group vs non respondeurs.

CONTACTS AND LOCATIONS:
Locations (1):
- Erasme Hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pees C, Glagau E, Hauser J, Michel-Behnke I. Reference values of aortic flow velocity integral in 1193 healthy infants, children, and adolescents to quickly estimate cardiac stroke volume. Pediatr Cardiol. 2013 Jun;34(5):1194-200. doi: 10.1007/s00246-012-0628-6. Epub 2013 Jan 24. PMID 23344893
- [Background] Wang J, Xu E, Xiao Y. Isotonic versus hypotonic maintenance IV fluids in hospitalized children: a meta-analysis. Pediatrics. 2014 Jan;133(1):105-13. doi: 10.1542/peds.2013-2041. Epub 2013 Dec 30. PMID 24379232
- [Background] Miller A, Mandeville J. Predicting and measuring fluid responsiveness with echocardiography. Echo Res Pract. 2016 Jun;3(2):G1-G12. doi: 10.1530/ERP-16-0008. Epub 2016 May 24. PMID 27249550
- [Background] Mercado P, Maizel J, Beyls C, Titeca-Beauport D, Joris M, Kontar L, Riviere A, Bonef O, Soupison T, Tribouilloy C, de Cagny B, Slama M. Transthoracic echocardiography: an accurate and precise method for estimating cardiac output in the critically ill patient. Crit Care. 2017 Jun 9;21(1):136. doi: 10.1186/s13054-017-1737-7. PMID 28595621
- [Background] Singh Y. Echocardiographic Evaluation of Hemodynamics in Neonates and Children. Front Pediatr. 2017 Sep 15;5:201. doi: 10.3389/fped.2017.00201. eCollection 2017. PMID 28966921
- [Background] Lopez L, Colan SD, Frommelt PC, Ensing GJ, Kendall K, Younoszai AK, Lai WW, Geva T. Recommendations for quantification methods during the performance of a pediatric echocardiogram: a report from the Pediatric Measurements Writing Group of the American Society of Echocardiography Pediatric and Congenital Heart Disease Council. J Am Soc Echocardiogr. 2010 May;23(5):465-95; quiz 576-7. doi: 10.1016/j.echo.2010.03.019. No abstract available. PMID 20451803
- [Background] Gaspar HA, Morhy SS. The Role of Focused Echocardiography in Pediatric Intensive Care: A Critical Appraisal. Biomed Res Int. 2015;2015:596451. doi: 10.1155/2015/596451. Epub 2015 Oct 28. PMID 26605333
- [Background] Lai WW, Geva T, Shirali GS, Frommelt PC, Humes RA, Brook MM, Pignatelli RH, Rychik J; Task Force of the Pediatric Council of the American Society of Echocardiography; Pediatric Council of the American Society of Echocardiography. Guidelines and standards for performance of a pediatric echocardiogram: a report from the Task Force of the Pediatric Council of the American Society of Echocardiography. J Am Soc Echocardiogr. 2006 Dec;19(12):1413-30. doi: 10.1016/j.echo.2006.09.001. No abstract available. PMID 17138024